CLINICAL TRIAL: NCT05339646
Title: A Phase I, Single and Multiple Dose, to Evaluate the Safety, Tolerability, and Pharmacokinetics of SSD8432 and SSD8432 Co-administrated in Healthy Adult Subjects
Brief Title: A Phase I Clinical Study of SSD8432 in Healthy Adult Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B02B11101-101
Record Dates: First submitted 2022-04-07; First posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Ritonavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- SSD8432 dose 1~7 (Experimental): Dose level 1 ~7 of SSD8432
  Interventions: Drug: SSD8432 dose 1~7 and Ritonavir
- SSD8432 dose 8~9 (Experimental): Dose level 8 ~9 of SSD8432
  Interventions: Drug: SSD8432 dose 8~9
- SSD8432 dose 10~12 (Experimental): Dose level 10 ~12 of SSD8432
  Interventions: Drug: SSD8432 dose 10~12 and ritonavir
- SSD8432 dose 13 (Experimental): Dose level 13 of SSD8432
  Interventions: Drug: SSD8432 dose 13 and Ritonavir
- SSD8432 dose 14 (Experimental): Dose level 14 of SSD8432
  Interventions: Drug: SSD8432 dose 14 and Ritonavir

INTERVENTIONS:
Drug: SSD8432 dose 1~7 and Ritonavir — Cohort 1 Period 1 single dose of SSD8432 dose 1 or placebo, on day 1. Period 2: single dose of SSD8432 dose 2 or placebo , on day 7. Period 3: single dose of SSD8432 dose 3 on day 13, ritonavir or placebo, before SSD8432 dose 3 and BID on SSD8432 dosing date
  Cohort 2:
  Period 1 single dose of SSD8432 dose 4 or placebo, on day 1 Period 2: single doses of SSD8432 dose 5 or placebo , on day 7 Period 3: single dose of SSD8432 dose 6 on day 13, ritonavir or placebo, before SSD8432 dose 3 and BID on SSD8432 dosing date
  Cohort 3:
  single dose of SSD8432 dose 7 or placebo on day1. ritonavir or placebo, before SSD8432 dose 7 and BID on SSD8432 dosing date.
  Arms: SSD8432 dose 1~7
Drug: SSD8432 dose 8~9 — Cohort 4: SSD8432 dose 8 or placebo, on day 1 ~day6. Cohort 5: SSD8432 dose 9 or placebo, on day 1 ~day6.
  Arms: SSD8432 dose 8~9
Drug: SSD8432 dose 10~12 and ritonavir — Cohort 6: SSD8432 dose 10 or placebo, on day 1 ~day6. Cohort 7: SSD8432 dose 11 or placebo, on day 1 ~day6. Cohort 8: SSD8432 dose 12 or placebo, on day 1 ~day6 Cohort 9: to be decided
  Arms: SSD8432 dose 10~12
Drug: SSD8432 dose 13 and Ritonavir — Cohort 10:
  Group A: SSD8432 dose 13, on day1 under fasting condition, on day 6 under fatty food condition, ritonavir, before SSD8432 dose 13 and BID on SSD8432 dosing date.
  Group B: SSD8432 dose 13, on day1 fatty food condition, on day 6 under fasting condition ,Ritonavir, before SSD8432 dose 13 and BID on SSD8432 dosing date
  Arms: SSD8432 dose 13
Drug: SSD8432 dose 14 and Ritonavir — Cohort 11: to be decided
  Arms: SSD8432 dose 14

SUMMARY:
This is a Phase I Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of SSD8432 in Healthy Adult Subjects

DETAILED DESCRIPTION:
108 healthy adult subjects (including 72 subjects in Part A to C, 16-24 subjects in Part D, and 8-12 subjects in optional Part E), including both males and females, will be enrolled in the phase I study.

This study will include Five parts: SSD8432 single dose and SSD8432 co-administrated with ritonavir (Part A), SSD8432 multiple dose (Part B), SSD8432 co-administrated with ritonavir multiple dose (Part C), SSD8432 co-administered ritonavir single dose in fasting and postprandial states (Part D: assessment of food effects) and optional part (Part E: Assessment of the safety and pharmacokinetics of SSD8432 in white healthy adult subjects)

ELIGIBILITY:
Inclusion Criteria:

* Male subjects' weight ≥ 50 kg, female subjects' weight ≥ 45 kg; body mass index ≥ 19 kg/m2 and ≤ 28 kg/m2.
* Female participants of child-bearing potential must agree to use adequate contraception from screening until 1 months after last dose.

Exclusion Criteria:

* History of any other acute or chronic illness (including cardiovascular, pulmonary, neurological, hepatic, rheumatic, hematological, metabolic or renal disorders), or use of medication that, in the opinion of the Principal Investigator, may not suitable for participating in this study.
* Subjects with a history of hematophobia or trypanophobia and unable to tolerate intravenous indwelling needle blood sampling.
* History of dysphagia or any other gastrointestinal disease possibly affecting drug absorption.
* Take special diet and cannot abide by the provided food and corresponding requirements in this study.
* Subject with a history of clinically significant hypersensitivity reactions to the active substance of SSD8432 or ritonavir or to any other components of drug products.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-04-07 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The Adverse events of SSD8432(Part A~D) | From signing ICF up to day 26
  Adverse events, including type, incidence, grade (determined with reference to NCI-CTCAE V5.0)
PK parameters(Part E) | Day 1 to Day 4
  Time for Cmax (Tmax)

SECONDARY OUTCOMES:
PK parameters(Part A~D) | Day 1 to Day 4
  Time for Cmax (Tmax)
The Adverse events of SSD8432(Part E) | From signing ICF up to day 26
  Adverse events, including type, incidence, grade (determined with reference to NCI-CTCAE V5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Yumei Yang, Study Director — Jiangsu Simcere Pharmaceutical Co., Ltd.
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yao B-F, Yang Y, Xu S-S, Tang B-H, Chen J, Guo Z-J, Hu H-L, Zhang W, Fu S-M, Zhang X-F, Hao G-X, Yang X-M, Song L-L, Ye P-P, Liu L, Zhu S-W, Zheng Y, Zhao W. Model-informed drug development in public health emergency of international concern: accelerating marketing authorization of simnotrelvir. Antimicrob Agents Chemother. 2025 Nov 5;69(11):e0061425. doi: 10.1128/aac.00614-25. Epub 2025 Sep 18. PMID 40965470
- [Derived] Yang XM, Yang Y, Yao BF, Ye PP, Xu Y, Peng SP, Yang YM, Shu P, Li PJ, Li S, Hu HL, Li Q, Song LL, Chen KG, Zhou HY, Zhang YH, Zhao FR, Tang BH, Zhang W, Zhang XF, Fu SM, Hao GX, Zheng Y, Shen JS, Xu YC, Jiang XR, Zhang LK, Tang RH, Zhao W. A first-in-human phase 1 study of simnotrelvir, a 3CL-like protease inhibitor for treatment of COVID-19, in healthy adult subjects. Eur J Pharm Sci. 2023 Dec 1;191:106598. doi: 10.1016/j.ejps.2023.106598. Epub 2023 Sep 30. PMID 37783378